CLINICAL TRIAL: NCT06352788
Title: From Opinion to Evidence: Multi-site Evaluation of Custom Dynamic Orthosis Best Practices
Acronym: AFOSVA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jason Wilken (Other)
Collaborators: Mayo Clinic (Other); Vanderbilt University Medical Center (Other); Navy Medical Center San Diego (U.S. Federal Agency); Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency); Johns Hopkins University (Other)
Responsible Party: Sponsor-Investigator, Jason Wilken, Associate Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 202007224; CDMRP-OP210038 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2024-04-02; First posted 2024-04-08 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: Foot Injury
Keywords: Ankle Foot Orthosis; Carbon Fiber; Gait; Biomechanics; Physical Performance
MeSH Terms: conditions — Foot Injuries

STUDY DESIGN:
Intervention Model Description: Participants will be cast and fit with either a carbon fiber custom dynamic orthosis (CDO) with a modular or mono design. After being fit with the CDO they will complete testing with the CDO in three different configurations (A, B, C) in a randomized order and without the CDO.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Study participants, investigators, and outcome assessors will be blinded to the condition being tested and will only be introduced to each condition as A, B, or C. Only study coordinators, who will verify adherence with the study protocol (CDO configuration), will not be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (6):
- NoCDO, A, B, C (Experimental): Participants will first be evaluated without a CDO (NoCDO), then in CDO configuration A, CDO configuration B, and finally CDO configuration C.
  Interventions: Device: Modular Carbon Fiber Custom Dynamic Orthosis (CDO); Device: Mono Carbon Fiber Custom Dynamic Orthosis (CDO)
- NoCDO, A, C, B (Experimental): Participants will first be evaluated without a CDO (NoCDO), then in CDO configuration A, CDO configuration C, and finally CDO configuration B.
  Interventions: Device: Modular Carbon Fiber Custom Dynamic Orthosis (CDO); Device: Mono Carbon Fiber Custom Dynamic Orthosis (CDO)
- NoCDO, B, A, C (Experimental): Participants will first be evaluated without a CDO (NoCDO), then in CDO configuration B, CDO configuration A, and finally CDO configuration C.
  Interventions: Device: Modular Carbon Fiber Custom Dynamic Orthosis (CDO); Device: Mono Carbon Fiber Custom Dynamic Orthosis (CDO)
- NoCDO, B, C, A (Experimental): Participants will first be evaluated without a CDO (NoCDO), then in CDO configuration B, CDO configuration C, and finally CDO configuration A.
  Interventions: Device: Modular Carbon Fiber Custom Dynamic Orthosis (CDO); Device: Mono Carbon Fiber Custom Dynamic Orthosis (CDO)
- NoCDO, C, A, B (Experimental): Participants will first be evaluated without a CDO (NoCDO), then in CDO configuration C, CDO configuration A, and finally CDO configuration B.
  Interventions: Device: Modular Carbon Fiber Custom Dynamic Orthosis (CDO); Device: Mono Carbon Fiber Custom Dynamic Orthosis (CDO)
- NoCDO, C, B, A (Experimental): Participants will first be evaluated without a CDO (NoCDO), then in CDO configuration C, CDO configuration B, and finally CDO configuration A.
  Interventions: Device: Modular Carbon Fiber Custom Dynamic Orthosis (CDO); Device: Mono Carbon Fiber Custom Dynamic Orthosis (CDO)

INTERVENTIONS:
Device: Modular Carbon Fiber Custom Dynamic Orthosis (CDO) — The CDO will use a modular design that includes a full length foot plate, a posterior carbon fiber strut, and a proximal cuff that wraps around the leg just below the knee.
  Other Names: Reaktiv (Fabtech Systems LLC, Everett WA)
Device: Mono Carbon Fiber Custom Dynamic Orthosis (CDO) — The CDO will use a mono design that includes a full length foot plate, a posterior carbon fiber strut, and a proximal cuff that wraps around the leg just below the knee.
  Other Names: Posterior Spring (Bio-Mechanical Composites, Inc., Des Moines, IA)

SUMMARY:
This study is designed to support evidence-based practice and optimal care by evaluating how different configurations of two types of carbon fiber custom dynamic orthoses (CDOs) influences outcomes following traumatic lower extremity injury.

DETAILED DESCRIPTION:
This study is designed to evaluate how different configurations of two types of carbon fiber custom dynamic orthoses (CDOs) influence outcomes following traumatic lower extremity injury. In this study, adult participants who still experiencing deficits including weakness and/or immobility more than two years post traumatic lower extremity injury will be randomized and fit with either modular or monolithic CDO.

Participants will then be evaluated without a CDO and with the CDO in three configurations in a randomized order: a proposed optimal benchmark configuration, a variation with the device in more dorsiflexion, and a variation with the device in greater plantarflexion. Multiple well-established tests will be used to compare outcomes between the different configurations.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 65
* 2 or more years from a traumatic injury below the knee
* Ability to be fit with an orthosis
* Any of the following:

  * Weakness of ankle plantarflexors (<4/5 on manual muscle test)
  * Limited pain-free ankle motion (dorsiflexion (DF) <10° or plantarflexion (PF) <20°)
  * Mechanical pain with loading to hindfoot/midfoot (>=4/10 Numerical pain rating scale)
  * Fusion or candidate for fusion of the ankle or hindfoot
  * Candidate for amputation secondary to ankle/foot injury and impairment

Exclusion Criteria:

* Pain greater than 8/10 at rest
* Ankle weakness or spasticity as a result of spinal cord injury or central nervous system pathology
* Use of an orthosis including the knee
* Non-ambulatory
* Surgery on study limb anticipated in next 4 months
* Medical or psychological conditions that would influence functional testing (e.g., severe traumatic brain injury, stroke, heart disease, vestibular disorder)
* Neurologic, musculoskeletal, or other conditions limiting function of the contralateral extremity
* Uncorrected visual or hearing impairments
* Pregnancy
* Non-English speaking
* BMI > 40

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-07-02 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
PROMIS Physical Function | Baseline
  The Patient Reported Outcome Information System (PROMIS) Physical Function Computer Adaptive Test (CAT) is a computerized assessment measuring physical function. It is scored using a T-score in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. In a given PROMIS domain, a T-score above 50 represents greater physical function than the population average. Larger scores are better.
PROMIS Pain Interference | Baseline
  The Patient Reported Outcome Information System (PROMIS) Pain Interference Computer Adaptive Test (CAT) is a computerized assessment measuring pain interference. It is scored using a T-score in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. In a given PROMIS domain, a T-score above 50 represents greater pain interference than the population average. Lower scores are better.
OPUS Satisfaction with Device and Services | Baseline
  Satisfaction with device and services will be assessed using the Orthotics Prosthetics Users' Survey Satisfaction With Device and Services Score (11-55). Lower scores indicate a better outcome and more satisfaction with the CDO and accompanying services.
Modified Socket Comfort Score - Comfort | Baseline
  Participants were asked to rate the comfort of each CDO configuration on a scale from 0-10 with 0 = most uncomfortable to 10 = most comfortable. Higher scores indicate more comfortable conditions, and are considered better.
Modified Socket Comfort Score - Smoothness | Baseline
  Participants were asked to rate the smoothness of each CDO configuration on a scale from 0-10 with 0 = most smooth to 10 = least smooth. Lower scores indicate smoother conditions, and are considered better.
Numerical Pain Rating Scale | Baseline
  Pain will be assessed using a standard 11-point numerical pain rating scale (NPRS), in which 0 = no pain and 10 = worst pain imaginable. Lower scores are considered better.
Preference - Ranked | Baseline
  The participant will be asked to rank order the conditions they have completed testing for at each visit: at the 3rd visit they will rank order their preference for using no orthosis or using the CDO in the first configuration, at the 4th visit they will rank order their preference for using no orthosis, using the CDO in the first configuration, and using the CDO in the second configuration, at the 5th visit they will rank order their preference for using no orthosis, using the CDO in the first configuration, using the CDO in the second configuration, and using the CDO in the third configuration.
Preference - CDO Configuration | Baseline
  For each CDO configuration, participants will be asked to rank their preference on a scale from 0 (least preferred) to 10 (most preferred) for a number of questions concerning CDO use. Higher scores indicate higher preferences and are considered better.
Four Square Step Test (seconds) | Baseline
  The 4SST (seconds) is a standardized timed test of balance and agility. Participants start in the lower left quadrant of a Maltese cross setting on the floor and are timed as they move counterclockwise (forward, right, backward, left) and then clockwise (right, forward, left, backward) around the cross. Participants are instructed to move as quickly as they safely can. Lower times indicate faster completion of the test and are considered better results.
Sit to Stand 5 Times (seconds) | Baseline
  STS5 (seconds) is a well-established timed measure of lower limb muscle strength and power. Participants are instructed to stand up and sit down 5 times as fast as possible. Lower scores indicate a faster time to complete the test and are considered better results.
Center of Pressure Velocity Magnitude (m/s) | Baseline
  The center of pressure (CoP) is the centroid of the forces acting on the foot during gait. The magnitude of the peak center of pressure velocity (m/s) is the fastest the CoP moves during gait.
Center of Pressure Velocity Timing (%stance) | Baseline
  The center of pressure (CoP) is the centroid of the forces acting on the foot during gait. The timing of the peak center of pressure velocity, is the percent of the stance phase (%stance) where the CoP is moving fastest during gait.
Ankle Zero Moment Crossing (%stance) | Baseline
  The ankle zero moment crossing is the point during the stance phase of gait (%stance) where the ankle moment transitions from a dorsiflexion to a plantarflexion moment.
Peak Ankle Dorsiflexion (degree) | Baseline
  Participants completed a biomechanical gait analysis session. Sagittal plane peak ankle joint dorsiflexion angle (degree) that occurs late in the stance phase of gait.
Peak Ankle Plantarflexion Moment (Nm/kg) | Baseline
  Participants completed a biomechanical gait analysis session. Sagittal plane peak ankle joint plantarflexion moment normalized to participant body weight (Nm/kg) that occurs late in the stance phase of gait.
Peak Ankle Push-Off Power (W/kg) | Baseline
  Participants completed a biomechanical gait analysis session. Sagittal plane peak ankle joint power normalized to body weight (W/kg) occurs late in the stance phase of gait.

SECONDARY OUTCOMES:
PROMIS Satisfaction with Participation in Social Activities | Baseline
  The Patient Reported Outcome Information System (PROMIS) satisfaction with participation in social activities Computer Adaptive Test (CAT) is a computerized assessment measuring satisfaction with participation in social activities. It is scored using a T-score in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. In a given PROMIS domain, a T-score above 50 represents greater participation in social activities than the population average, larger scores are considered better.
PROMIS Satisfaction with Participation in Discretionary Social Activities | Baseline
  The Patient Reported Outcome Information System (PROMIS) satisfaction with participation in social activities Computer Adaptive Test (CAT) is a computerized assessment measuring satisfaction with participation in social activities. It is scored using a T-score in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. In a given PROMIS domain, a T-score above 50 represents greater participation in discretionary social activities than the population average, larger scores are considered better.
PROMIS Depression | Baseline
  The Patient Reported Outcome Information System (PROMIS) depression Computer Adaptive Test (CAT) is a computerized assessment measuring depression. It is scored using a T-score in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. In a given PROMIS domain, a T-score above 50 represents greater levels of depression than the population average, lower scores are considered better.

OTHER OUTCOMES:
Ankle Range of Motion (degrees) | Baseline
  Participants completed a biomechanical gait analysis session. Sagittal plane ankle range of motion (degrees) was measured throughout the gait cycle. Smaller range of motion is expected with each CDO.

CONTACTS AND LOCATIONS:
Overall Officials: Jason M Wilken, PT, PhD, Principal Investigator — University of Iowa
Locations (5):
- United States (5):
  - Naval Medical Center San Diego - Clinical Biomechanics Laboratory, San Diego, California
  - University of Iowa, Iowa City, Iowa
  - Minneapolis VA Health Care System - Motion Analysis Laboratory, Minneapolis, Minnesota
  - Mayo Clinic - Motion Analysis Lab, Rochester, Minnesota
  - Vanderbilt University - Zelik Lab For Biomechanics & Assistive Technology, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No